CLINICAL TRIAL: NCT06610045
Title: The Burden of Multiple Myeloma on Patients and Caregivers Quality of Life: a Canadian Real-World Study
Status: Completed | Type: Observational
Sponsor: PeriPharm (Other)
Responsible Party: Sponsor
Other Study IDs: PROxy202301
Record Dates: First submitted 2024-09-12; First posted 2024-09-24 (Actual); Last update posted 2025-03-13 (Actual); Status verified 2025-03

CONDITIONS: Multiple Myeloma; Caregiver Subjective Burden; Quality of Life (QOL)
Keywords: quality of life; real-world; observational; myeloma; caregiver
MeSH Terms: conditions — Multiple Myeloma; Neoplasms, Plasma Cell

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Patients with multiple myeloma: Patients with multiple myeloma member of Myeloma Canada database
  Interventions: Other: No intervention
- Caregivers of patients with myeloma: Caregiver of a multiple myeloma patient member of Myeloma Canada database
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — No specific intervention is assess in this study.

SUMMARY:
The purpose of this observational study is to estimate the burden of multiple myeloma on patients and caregivers in terms of QoL. Additionally, this study will assess the correlation between QoL, obtained from commonly used and validated questionnaires, and the perceptions of both patients and caregivers respectively., obtain from a 10-point scale and a comment box.

DETAILED DESCRIPTION:
Potential participants will be identified by Myeloma Canada using their database. Myeloma Canada is a registered non-profit organization created by, and for, Canadians impacted by multiple myeloma. As part of Myeloma Canada website, patients and caregivers can subscribe to a mailing list to receive their monthly newsletter and to participate in surveys. This database comprises about 5,000 individuals, including patients and caregivers.

An e-mail will be sent to 600 patients and 200 caregivers randomly selected to invited them to participate in the survey. Interested participants will be invited to visit the Participant Portal on the PROxy website (https://periproxy.com/en), to sign the informed consent form and complete online questionnaires. Upon request, paper-based documents (i.e., informed consent form and questionnaires) can also be sent by mail. The following questionnaires will be used:

Patients

* Patient Information Questionnaire (i.e., baseline characteristics)
* EORTC QLQ-C30
* EORTC QLQ-MY20
* EQ-5D-5L
* ESAS-R
* Patients Perspective

Caregivers

* Caregiver Information Questionnaire (i.e., baseline characteristics)
* CarGOQoL
* Caregivers Perspective

If the sample size (i.e., 300 patients and 100 caregivers) is not reached one month after the first e-mail, an invitation e-mail will be sent to an additional 600 eligible patients and/or 200 caregivers randomly selected. This scheme of participant identification will be performed until the sample size is reached.

ELIGIBILITY:
Inclusion Criteria:

1. 18 years of age or older;
2. Part of the Myeloma Canada database;

   1. Identified as a patient with MM or
   2. Identified as a current caregiver of a patient with MM at the time of participation.
3. Ability to read and understand English or French;
4. Signature of informed consent form (ICF).

Exclusion Criteria:

No exclusion criteria

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with myeloma and caregivers of patients with myeloma who are part of Myeloma Canada database
Sampling Method: Non-Probability Sample
Enrollment: 400 (Actual)
Dates: Start 2024-10-15 (Actual); Primary Completion 2025-02-24 (Actual); Study Completion 2025-03-12 (Actual)

PRIMARY OUTCOMES:
To estimate quality of life of patients with myeloma and caregivers of patients with myeloma | From enrollment until sample size is reached

SECONDARY OUTCOMES:
To assess the correlation between QoL scores and perception of patients and caregivers respectively | From recruitment until sample size is reached

CONTACTS AND LOCATIONS:
Locations (1):
- PROxy Network, an initiative of PeriPharm inc., Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No